CLINICAL TRIAL: NCT00867009
Title: A Phase 2 Study of Pemetrexed and Cisplatin Plus Cetuximab Followed by Pemetrexed and Cetuximab Maintenance Therapy in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (Stage IIIB or IV) Other Than Predominantly Squamous Cell Histology
Brief Title: A Study of Induction and Maintenance Treatment of Advanced or Metastatic Non Squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10726; H3E-MC-S104 (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2012-05-16 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2014-09

CONDITIONS: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Cisplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Induction/maintenance Therapy (Experimental): pemetrexed, cisplatin and cetuximab followed by pemetrexed and cetuximab
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Cetuximab

INTERVENTIONS:
Drug: Pemetrexed — Induction therapy: 500 mg/m², intravenous, on Day 1 of each 21-day cycle for 4 to 6 cycles Maintenance therapy: 500 mg/m², intravenous, on Day 1 of each 21-day cycle until progressive disease or treatment discontinuation
  Other Names: Alimta; LY231514
Drug: Cisplatin — Induction therapy: 75 mg/m², intravenous, on Day 1 of each 21-day cycle for 4 to 6 cycles
Drug: Cetuximab — Induction therapy: Loading dose of 400 mg/m², intravenous, on Day 1 of cycle 1, then 250 mg/m², intravenous, weekly for 4 to 6 cycles, 21 day cycles
  Maintenance therapy: 250 mg/m², intravenous, weekly until progressive disease or treatment discontinuation

SUMMARY:
This study will estimate the response rate in patients with advanced or metastatic non-squamous Non-Small Cell Lung Cancer. Patients who don't progress after 4 to 6 cycles of induction treatment with pemetrexed, cisplatin and cetuximab will receive maintenance treatment with pemetrexed and cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Patient must sign an informed consent document for clinical and translational research.
* Patient must have locally advanced or metastatic nonsquamous Non-Small Cell Lung Cancer.
* Patient must have biological tissue available from your diagnosis tumor for detection of some biomarkers (translational research).
* Patient cannot be receiving nor have received any prior systemic anticancer therapy, immunotherapy, targeted therapy, or biological therapy for your lung cancer (except chemotherapy given after surgery if it has been completed more than one year before the study entry).
* Patient is allowed to have had prior radiation therapy as long as it was not more than 25% of the bone marrow and did not include the whole pelvis. Prior radiation therapy should be completed at least 2 weeks prior to first study drug. Thoracic radiation must be completed more than 12 weeks before the study entry. You must be recovered from the toxic effects.
* Patient must have at least 1 measurable tumor lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines.
* Patient must at least be able to be physically mobile, take care of yourself, and must be up and about and able to perform light activities such as light housework or office work.
* Test results assessing the function of blood forming tissue, kidneys, and liver must be satisfactory.
* Females must be sterile, postmenopausal or on contraception.
* Males must be on contraception or sterile (for example post-vasectomy).

Exclusion Criteria:

* Patient cannot have symptomatic central nervous system metastases.
* Patient cannot have an active infection or other serious condition that your doctor thinks would make you unable to participate.
* Patient cannot have a serious cardiac condition, such as a heart attack, angina, or heart disease within 6 months of entering the trial.
* Patient cannot have had a another form of cancer other than superficial basal cell and superficial squamous (skin) cell cancer, or carcinoma in situ of the cervix within the last 5 years.
* Patient cannot have had significant neurologic or psychiatric disorders including dementia, seizures and bipolar disorder.
* Patient cannot have moderate or severe peripheral neuropathy
* Patient cannot have received treatment within 30 days with any experimental drug.
* Patient cannot have had a major surgery within the last 4 weeks.
* Patient cannot have previously received treatment with transduction inhibitors or Epidermal Growth Factor Receptor (EGFR)-targeting therapy.
* Patient cannot have prior known allergic/hypersensitivity reaction to any of the components of study treatments.
* Females cannot be pregnant or breastfeeding.
* Patient is unable to stop taking more than 1.3 grams of aspirin on a daily basis or other aspirin like medication (non-steroidal antiinflammatory drugs: NSAIDs) for a few days during each cycle of therapy.
* Patient is unable or unwilling to take folic acid, injections of vitamin B12, or corticosteroids.
* Patient cannot have fluid around your lungs or in your abdomen (pleural effusions or ascites) that cannot be controlled by drainage or other procedures.
* Patient cannot have received a yellow fever vaccination within the previous 30 days or plan to have it.
* Patient cannot have known drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2009-04; Primary Completion 2011-05 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (24):
- Austria (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salzburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wels
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Halle
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Homburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mannheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
- Greece (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
- Italy (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palermo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Potenza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Treviso
- Netherlands (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., 's-Hertogenbosch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Groningen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Maastricht
- Spain (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lleida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reus

RESULTS

PARTICIPANT FLOW:
Groups:
- Pem/Cis + Cet: Induction Therapy: 500 mg/m² pemetrexed (Pem)on Day 1 of every 21-day cycle, 75 mg/m² cisplatin (Cis) on Day 1 of every 21-day cycle and 400 mg/m² cetuximab (Cet) given intravenously (IV) on Day 1 of Cycle 1 and 250 mg/m² once weekly thereafter. Induction period is 4 to 6 cycles.
  Maintenance Therapy: 500 mg/m² pemetrexed (Pem) given intravenously (IV) on Day 1 of each 21 day cycle and 250 mg/m² cetuximab (Cet) given weekly until progressive disease (PD) or treatment discontinuation.
Period: Induction Period
Arm/Group | Pem/Cis + Cet
Started | 113 (Participants with Stage IIIB/IV non-squamous (NS) non-small cell lung cancer (NSCLC))
Received at Least 1 Dose of Study Drug | 113
Protocol Qualified (PQ) Population | 109 (Stage IIIB/IV NS-NSCLC, no concurrent chemotherapy, measurable disease, ≥1 dose study drug.)
Completed | 51 (Participants continued on the study in the Maintenance Period.)
Not Completed | 62
Not completed — Nonserious Adverse Event | 5
Not completed — Serious Adverse Event | 10
Not completed — Death due to serious adverse event | 6
Not completed — Death due to Study Disease | 4
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 8
Not completed — Physician Decision | 3
Not completed — Progressive Disease (PD) | 25
Period: Maintenance Period
Arm/Group | Pem/Cis + Cet
Started | 51
Completed | 47 (Participant was considered completed if they had PD, death, or stopped receiving study drug.)
Not Completed | 4
Not completed — On-going in the Study at Data Cut-off | 4

BASELINE CHARACTERISTICS:
Arm/Group | Pem/Cis + Cet
Number analyzed (Participants) | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.15 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 72
Race/Ethnicity, Customized [Number; unit: participants]
  White | 113
Region of Enrollment [Number; unit: participants]
  Greece | 12
  Spain | 25
  Austria | 6
  Germany | 28
  Netherlands | 16
  Italy | 26
Eastern Co-operative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. ECOG Performance Score: 0 - Fully Active; 1 - Ambulatory, Restricted Strenuous Activity; 2 - Ambulatory, No Work Activities; 3 - Partially Confined to Bed, Limited Self Care; 4 - Completely Disabled; 5 - Death
  participants
    0 - Fully Active | 56
    1 - Ambulatory, Restricted Strenuous Activity | 57
Disease Stage [Number; unit: participants] — Stage means how big the tumor is and how far it has spread. Stages range from 0 (not spread) to IV (spread throughout the body). Stage IIIB - the cancer has spread to nearby tissue or spread to far away lymph nodes. Stage IV - the cancer has spread to other organs of the body such as the other lung, brain, or liver
  participants
    Stage IIIB | 9
    Stage IV | 104
Pathological Diagnosis [Number; unit: participants]
  Adenocarcinoma (Adeno), Breast | 1
  Carcinoma, Adenosquamous,Lung, Predominantly Adeno | 1
  Large Cells Lung Carcinoma | 5
  Malignant Neoplasm, Adeno Lung | 88
  Non-Small Cell Lung (NSCL) Cancer | 9
  Poorly Differentiated Non-Small Cell | 8
  Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Tumor Response (Objective Tumor Response Rate)
Description: Response was assessed using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response (CR)=disappearance of all target lesions; Partial Response (PR)=30% decrease in sum of longest diameter of target lesions. Tumor response is presented as a percentage (%) and is the number of participants with a CR plus PR divided by the number of participants in the protocol qualified (PQ) population, then multiplied by 100.
Time Frame: From start of treatment until documented best response. (up to 18.9 months)
Population: Outcome measure was assessed using the Protocol Qualified (PQ) population.
Measure: Number; unit: percentage of participants
Arm/Group | Pem/Cis + Cet
Number analyzed (Participants) | 109
percentage of participants | 38.5
Statistical Analysis 1: Comparison: Pem/Cis + Cet; Test type: Superiority or Other; Percentage of participants with response = 38.5, 80% CI 2-sided [32.30 to 45.09]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is measured from study entry until disease progression, death or date of last contact. Progressive disease (PD) was determined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. PD = 20% increase in sum of longest diameter of target lesions or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. For participants not known to have died or have had objective PD as of the data cutoff date, PFS was censored at the date of the last objective progression-free disease assessment.
Time Frame: From start of treatment until documented disease progression or death from any cause (up to 18.9 months)
Population: Outcome measure was assessed using the Protocol Qualified (PQ) population.
Measure: Median (Full Range); unit: months
Arm/Group | Pem/Cis + Cet
Number analyzed (Participants) | 109
months | 5.82 [0.03 to 18.89]
Statistical Analysis 1: Comparison: Pem/Cis + Cet; Test type: Superiority or Other; Median number of months = 5.82, 80% CI 2-sided [4.40 to 6.70]

3. Secondary Outcome: The Percentage of Participants Still Living at One Year (One Year Survival Rate)
Description: The one year survival rate is presented as percentage (%) of participants still living at one year and is the number of participants that are still alive at one year divided by the number of participants in the protocol qualified (PQ) population, which is then multiplied by 100.
Time Frame: One year
Population: Outcome measure was assessed using the Protocol Qualified (PQ) population.
Measure: Number; unit: percentage of participants
Arm/Group | Pem/Cis + Cet
Number analyzed (Participants) | 109
percentage of participants | 45
Statistical Analysis 1: Comparison: Pem/Cis + Cet; Test type: Superiority or Other; Percentage of participants with response = 45, 80% CI 2-sided [39 to 51]

4. Secondary Outcome: The Percentage of Participants With Complete Response (CR), Partial Response (PR) or Stable Disease (SD) (Disease Control Rate [DCR])
Description: The DCR is presented as percentage (%) and is the number of participants with a best tumor response of CR, PR, or SD divided by the number of participants in the protocol qualified (PQ) population, then multiplied by 100. Best tumor response of CR, PR, or SD was determined from the sequence of tumor response assessments. Tumor response was assessed using RECIST criteria. CR=disappearance of all target lesions; PR=30% decrease in sum of longest diameter of target lesions; SD=small changes that do not meet above criteria.
Time Frame: From start of treatment until documented best tumor response (up to 18.9 months)
Population: Outcome measure was assessed using the Protocol Qualified (PQ) population.
Measure: Number; unit: percentage of participants
Arm/Group | Pem/Cis + Cet
Number analyzed (Participants) | 109
percentage of participants | 59.6
Statistical Analysis 1: Comparison: Pem/Cis + Cet; Test type: Superiority or Other; Percentage of participants with response = 59.6, 80% CI 2-sided [53.06 to 65.94]

ADVERSE EVENTS:
Description: Serious Adverse Events are presented regardless of causality.
Arm/Group | Pem/Cis + Cet
Serious Adverse Events (participants affected / at risk) | 61/113
Other Adverse Events (participants affected / at risk) | 101/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pem/Cis + Cet (N=113)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (7)
Atrial flutter (Cardiac disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Diplopia (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Diverticular perforation (Gastrointestinal disorders) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Device occlusion (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (3)
General physical health deterioration (General disorders) | 3 (4)
Malaise (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (3)
Obstruction (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (3)
Sudden death (General disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Biliary sepsis (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 2 (2)
Gangrene (Infections and infestations) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Peritonitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Uterine haemorrhage (Reproductive system and breast disorders) | 1/41 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Peripheral ischaemia (Vascular disorders) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Pem/Cis + Cet (N=113)
Anaemia (Blood and lymphatic system disorders) | 20 (38)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Haemoglobinaemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 24 (60)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 25 (72)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (9)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac fibrillation (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (2)
Deafness (Ear and labyrinth disorders) | 4 (5)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 5 (5)
Vertigo (Ear and labyrinth disorders) | 2 (3)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1)
Blepharitis (Eye disorders) | 3 (3)
Diplopia (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 5 (5)
Eye oedema (Eye disorders) | 1 (1)
Eyelid disorder (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 10 (12)
Ocular hyperaemia (Eye disorders) | 1 (1)
Ocular surface disease (Eye disorders) | 2 (2)
Ulcerative keratitis (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 7 (8)
Abdominal pain upper (Gastrointestinal disorders) | 5 (8)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 29 (33)
Diarrhoea (Gastrointestinal disorders) | 24 (36)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 8 (9)
Eructation (Gastrointestinal disorders) | 2 (2)
Gastritis (Gastrointestinal disorders) | 6 (9)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 (1)
Glossitis (Gastrointestinal disorders) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 51 (95)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 2 (3)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 23 (38)
Vomiting (Gastrointestinal disorders) | 34 (58)
Asthenia (General disorders) | 15 (20)
Catheter site pain (General disorders) | 1 (1)
Chest pain (General disorders) | 8 (8)
Chills (General disorders) | 1 (1)
Extravasation (General disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 37 (81)
Feeling cold (General disorders) | 2 (2)
Generalised oedema (General disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Localised oedema (General disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Mucosal dryness (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 21 (30)
Oedema peripheral (General disorders) | 9 (12)
Pain (General disorders) | 2 (2)
Peripheral swelling (General disorders) | 1 (1)
Pyrexia (General disorders) | 14 (19)
Ulcer (General disorders) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (2)
Contrast media allergy (Immune system disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 3 (4)
Seasonal allergy (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 16 (25)
Cystitis (Infections and infestations) | 2 (2)
Ear infection (Infections and infestations) | 1 (1)
Eye infection (Infections and infestations) | 2 (2)
Folliculitis (Infections and infestations) | 5 (5)
Gastroenteritis (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Nail bed infection (Infections and infestations) | 1 (1)
Nail infection (Infections and infestations) | 5 (6)
Nasopharyngitis (Infections and infestations) | 4 (4)
Oral candidiasis (Infections and infestations) | 1 (1)
Oral fungal infection (Infections and infestations) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 2 (2)
Penile infection (Infections and infestations) | 1/72 (3)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 4 (5)
Rhinitis (Infections and infestations) | 2 (3)
Sinusitis (Infections and infestations) | 2 (3)
Skin infection (Infections and infestations) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1)
Upper aerodigestive tract infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (5)
Vaginal infection (Infections and infestations) | 2/41 (2)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Radiation skin injury (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Vascular injury (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (13)
Aspartate aminotransferase increased (Investigations) | 4 (17)
Blood calcium (Investigations) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1)
Blood creatinine decreased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 5 (8)
Blood magnesium decreased (Investigations) | 4 (6)
Blood potassium decreased (Investigations) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (6)
Glomerular filtration rate decreased (Investigations) | 1 (1)
Haemoglobin (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 11 (20)
Neutrophil count decreased (Investigations) | 3 (4)
Platelet count decreased (Investigations) | 6 (8)
Protein c increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 11 (11)
Weight increased (Investigations) | 1 (2)
White blood cell count decreased (Investigations) | 3 (5)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 21 (34)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 5 (8)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 8 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (19)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (13)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/41 (1)
Ageusia (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 15 (15)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 8 (9)
Headache (Nervous system disorders) | 9 (15)
Hypogeusia (Nervous system disorders) | 1 (2)
Neuralgia (Nervous system disorders) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 3 (3)
Paraesthesia (Nervous system disorders) | 3 (4)
Paraparesis (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 12 (14)
Presyncope (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 4 (4)
Depression (Psychiatric disorders) | 3 (4)
Fear (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5)
Sleep disorder (Psychiatric disorders) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2)
Renal colic (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 1/72 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1/72 (1)
Menstruation irregular (Reproductive system and breast disorders) | 1/41 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1/41 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (24)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (28)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (10)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (12)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (4)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 2 (2)
Intertrigo (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 6 (7)
Nail toxicity (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 62 (88)
Rash follicular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (2)
Catheter placement (Surgical and medical procedures) | 1 (1)
Dental implantation (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (5)
Hypotension (Vascular disorders) | 3 (4)
Phlebitis (Vascular disorders) | 1 (1)
Phlebitis superficial (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days